CLINICAL TRIAL: NCT06054581
Title: A Study of Animal Bite Among Victims Seeking Medical Services at the Concerned Hospitals in Assiut City
Brief Title: Animal Bite Victims Seeking Medical Services at Concerned Hospitals
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, alyaa abdelaal mohamed abdelaal, assisstant lecturer, Assiut University
Other Study IDs: animal bite
Record Dates: First submitted 2023-09-20; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Vaccine-Preventable Diseases
Keywords: animal bite, vaccine compliance
MeSH Terms: conditions — Vaccine-Preventable Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: health seeking behavior — health seeking behavior in the form of wound management and receving anti rabies immunization

SUMMARY:
The goal of this observational study is to study the magnitude of the animal bite problem during one year ,to determine the percentage of compliance for full PEP doses and factors affecting the health seeking behavior among these victims.

To assess the management of the wound (first aid management done by the patient and in the hospital).

Participants will be asked to answer a questionnaire consisting of five parts and followed for completing their anti-rabies vaccination schedule.

DETAILED DESCRIPTION:
Animal bites pose a major public health problem in children and adults worldwide. Numerous animal species have the potential to bite humans leading to rabies which is a disease of mammals , including dogs, wolves, foxes, cats, lions, mongooses, bats, monkeys and humans, However, the use of dogs as pets or companions, and for security, hunting, and breeding has contributed to their growing population.

Surveillance data revealed that people in Egypt experience a large number of animal bites annually with more than 200,000 animal bites recorded each year mostly from dogs. On average 60 people die annually from rabies in Egypt.

Rabies is 100% fatal disease but can be prevented with successful rabies control program which comprise of three pillars:1. Community participation; education, public awareness. 2. Access to mass vaccination of dogs. 3. Access to post bite treatment.

PEP is the administration of wound care and immunization after potential exposure to the rabies virus.

As a part of zero by 30 strategy set by WHO to control dog-mediated human rabies by 2030, the strategic advisory group of experts of the WHO needed the current scenario of health-seeking behavior of exposed individuals and the use of rabies vaccines and immunoglobulin in rabies endemic countries. In this regard, perception of victims and their attitude towards treatment forms an important role for prevention against rabies. It is also necessary to detect trends to evaluate the effect of preventive efforts implemented by the Ministry of Health.

ELIGIBILITY:
Inclusion Criteria:

* victims recently exposed to bite by any animal causing rabies

Exclusion Criteria:

* other types of animal bites

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: victims who recently exposed to animal bite attending to receive their first vaccination dose
Sampling Method: Non-Probability Sample
Enrollment: 662 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
anti-rabies vaccination compliance among animal bite victims | each patient will be followed for 2 months after the first visit till completing the required sample
  follow up of victims coming to receive their vaccination for the first time

CONTACTS AND LOCATIONS:
Overall Officials: alyaa abdelaal, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kenu E, Ganu V, Noora CL, Adanu R, Lartey M. Management of dog bites by frontline service providers in primary healthcare facilities in the Greater Accra Region of Ghana, 2014-2015. Infect Dis Poverty. 2018 Feb 28;7(1):18. doi: 10.1186/s40249-018-0398-3. PMID 29502522
- [Result] Jakasania AH, Mansuri FM, Dixit GT. An association of knowledge and misconceptions with health seeking behaviour for dog bite: a cross-sectional study in Ahmedabad. Int J Comm Med Public Heal. 2017 Jun 23;4(7):2592-5.
- See also: WHO. Animal bites [Internet]. 2018 [cited 2023 May 17] — https://www.who.int/news-room/fact-sheets/detail/animal-bites